CLINICAL TRIAL: NCT05118919
Title: A Randomised Placebo-controlled Safety Study of Lactobacillus Reuteri BGP-014 in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: A Safety Study of Lactobacillus Reuteri BGP-014 in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioGaia Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUCH-1
Record Dates: First submitted 2021-10-26; First posted 2021-11-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental)
  Interventions: Biological: BGP-014
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BGP-014 — Oral capsule containing lyophilised Lactobacillus reuteri
  Arms: Active
Biological: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability and preliminary efficacy of Lactobacillus reuteri BGP-014 in mild to moderate active Ulcerative Colitis (UC) patients as an oral administered local treatment in addition to Standard of Care (SoC) treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study.
* Diagnosed previously with UC (> 6 months earlier) determined by clinical and endoscopic histopathology (pathology showing chronic inflammatory changes). ≥1 documented previous flare-up and with last resolved flare >3 months away.
* Active UC determined by sigmoidoscopy before randomisation of study (baseline) and defined as a total Mayo index score of 4 to 10 points (endoscopic subscore ≥1, rectal bleeding ≥1).
* Permitted concomitant SoC medications include: Oral aminosalicylates (5-ASA), with a stable dose (1.6-4.8g/ day) for at least 12 days prior to screening, Visit 1. Steroids (dose ≤15mg at screening, Visit 1) with further tapering of dose in accordance with SoC until steroid tx termination. Immunomodulator, as: 6-Mercaptopurine, Azathioprine, Methotrexate (Stable dose for > 12 weeks prior to screening, Visit 1).
* Females of childbearing potential must use effective contraceptives

Exclusion Criteria:

1. Involvement in any investigational drug or device study within 30 days prior to this study
2. Known intolerance of 5-ASA or sulphasalazine medications
3. Biologics or FMT treatment less than 12 weeks before screening
4. No 5-ASA or steroid topical treatment is allowed
5. Antibiotic treatment < 1 month prior the study
6. Unable to maintain stable dose of NSAIDs and PPIs
7. Evidence of on-going extensive colitis
8. Fever, defined as a temperature of >38.5 °C, at Visit 1
9. Anaemia, Hb value below 100
10. Evidence of on-going toxic megacolon
11. Presence of obstructive diseases of the gastrointestinal system
12. Any clinically significant concomitant disease that might interfere with patient safety
13. Unwilling to withdraw probiotic supplements. Yoghurts without supplemented bacteria are permitted
14. Pregnant
15. Planned abdominal surgery
16. Judged unable by the physician to comprehend information regarding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Up to 10 weeks
  The primary objective is to evaluate the safety and tolerability of BGP-014.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellström, Professor, Principal Investigator — Uppsala University Hospital
Locations (4):
- Sweden (4):
  - Department of Gastroenterology and Hepatology, Linköping University Hospital, Linköping
  - Gastroenterology Department, Danderyds Hospital, Stockholm
  - Gastroenterology Department, Ersta Hospital, Stockholm
  - Department of Medical Sciences Gastroenterology and Hepatology, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No